CLINICAL TRIAL: NCT05378308
Title: Outcomes regiStry for Non-vitamin k Antagonist Oral anticoagUlants treatmeNt in variouS tHrombotIc dIseases for Better cliNical practicE (SUNSHINE)
Brief Title: NOACs Use in AF or VTE (SUNSHINE Registry)
Status: Recruiting | Type: Observational
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0508
Record Dates: First submitted 2022-05-08; First posted 2022-05-18 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation; Venous Thromboembolism; Oral Anticoagulant
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with Atrial Fibrillation (AF) or venous thromboembolism (VTE) — Patients with AF or VTE; OAC treatment patterns according to patient demographics, clinical factors, risk stratification, geographic regions, local NOAC medical insurance policy and NOACs availability

SUMMARY:
The outcomes regiStry for non-vitamin k antagonist oral anticoagUlants treatmeNt in variouS tHrombotIc dIseases for better cliNical practicE (SUNSHINE) is a multicenter, prospective, observational non-interventional inpatient/outpatient disease registry to assess the utilization of Non-vitamin k antagonist oral anticoagulants (NOACs), and associated outcomes. The SUNSHINE registry will focus on the collection and analysis of observational data in medical records from hospital information system (HIS) to evaluate the outcomes related with these NOACs when applied in extensive patient populations outside of clinical research studies. The registry will also allow for mainly combining the atrial fibrillation (AF) and venous thromboembolism (VTE) databases. In brief, the SUNSHINE registry will provide important information on the outcomes of NOACs in routine practice and gather further information on its safety and effectiveness.

DETAILED DESCRIPTION:
The SUNSHINE registry will generate the extensive integrated repository of routine clinical care data for NOACs use in patients for various clinical scenarios (mainly with AF or VTE). It will provide important information on the use of NOACs in routine clinical care and gather further information on its safety and effectiveness. The study will compare the characteristics of patients newly anticoagulated with either VKAs or NOACs, to describe the reasons for discontinuing the previous anticoagulant strategy and/or choosing the newly initiated anticoagulant treatment, and to precisely describe the prescriptions of patients newly initiated with a NOAC agent, the treatment patterns, clinical course and the clinical outcomes related with their use. The registry will be a multicenter-collaborated study led by clinical pharmacists and cooperate with health care providers (eg, cardiologists, internists, electrophysiologists, general practitioners, and so on). Target enrollment will be approximately 5,000 patients. It is expected that enrollment will finish in approximately 5 years. Patients who meet the eligibility criteria will be included. Approval from the Henan Provincial People's Hospital Institutional Review Board will be obtained before starting the survey. Since the sensitive data of each patient will be removed (e.g., by name and identification), and only presented in aggregate; therefore, informed consent is waived for this study. Confidentiality will be ensured in accordance with the Declaration of Helsinki. Data collection will include patients' electronic medical records (include demographics, clinical characteristics, medical management, laboratory measurements and imaging parameters, prescription information), the catigories of treating physicians, local NOAC medical insurance policy and NOACs availability of each institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically diagnosed with AF (eg, by electrocardiogram, Holter monitoring, implanted device, etc) or VTE (initial or recurrent acute VTE)
* Patients who use OACs therapy (including NOAC or VKA) within the preceding 3 months
* Patients can be enrolled from both inpatient or outpatient settings

Exclusion Criteria:

* AF resulting from reversible cause factors (e.g., thyroid disease, postoperative AF)
* Patients with a diagnosis of valvular AF (valvular AF mainly refers to patients with AF that have either rheumatic valvular disease [predominantly mitral stenosis] or mechanical heart valves)
* Patients participating in an ongoing clinical trial in AF or VTE
* Have Multiple anticoagulation indications apart from AF or VTE
* Patients with incomplete information (illogical data, missing or insufficient data)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NOACs use in patients for various clinical scenarios (mainly with AF or VTE).
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Profiles of patients with OACs | During hospitalization
  Patient's characteristics such as age, gender, weight, BMI, disease status; disease characteristics like co-morbidities (congestive heart failure history, hypertension, diabetes mellitus, stroke/transient ischemic attack)/thromboembolism history, vascular disease history, renal impairment, liver impairment, prior major bleeding), treatment history (previous anticoagulation strategy, duration and indication of previous anticoagulation treatment).
Patients with AF prescribed with OAC | During hospitalization
  Difference in the proportion of patients with AF prescribed with OAC between the appropriate use and the inappropriate use group.
Patients with VTE prescribed with OAC | During hospitalization
  Difference in the proportion of patients with VTE prescribed with OAC between the appropriate use and the inappropriate use group.

SECONDARY OUTCOMES:
Number of major bleeding events | 5 years
  Major bleeding will be defined according to International Society of Thrombosis and Hemostasis (ISTH) criteria.
Number of adverse cardiac events | 5 years
  Cardiac events are defined as stroke or non-central nervous system (non-CNS) systemic embolism, myocardial infarction, and cardiovascular death.

CONTACTS AND LOCATIONS:
Overall Officials: Shujuan Zhao, Study Director — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China